CLINICAL TRIAL: NCT05880875
Title: Enhancing Early Care and Education Through Reflective Supervision to Promote Adaptive Emotion Regulation in Young Children
Brief Title: Enhancing Early Care and Education Through Reflective Supervision
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Bradley Hospital (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Lindsay Huffhines, PhD, Research Scientist, Bradley Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: K23HD107243 (NIH); K23HD107243 (NIH)
Record Dates: First submitted 2023-05-18; First posted 2023-05-30 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Emotion Regulation
Keywords: Reflective Supervision; Reflective Capacity; Early Care and Education; Social-Emotional Development
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Intervention Model Description: Participants (i.e., early learning supervisors) will be randomized to the experimental condition (i.e., the Reflective Supervision enhancement) or the waitlist control condition (i.e., business-as-usual).
Who Masked: Outcomes Assessor
Masking Description: Classroom observations will be conducted by study staff who are not aware of which study condition (i.e., experimental or waitlist control) participants are enrolled in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reflective Supervision Enhancement (Experimental): The Reflective Supervision enhancement is a professional development series for supervisors of state pre-kindergarten programs that is designed to build skills in using Reflective Supervision with teachers. The goal of the Reflective Supervision enhancement is to provide supervisors with foundational knowledge in Reflective Practice and Supervision and increase their use of Reflective Supervision principles and practices within their work. The series consists of a day-long foundational training and nine skills-focused workshops. Supervisors are expected to receive 8 hours of foundational training prior to the start of the academic year, and nine 2-hour monthly small groups over the course of the academic year.
  Interventions: Behavioral: Reflective Supervision Enhancement
- Business-As-Usual Waitlist Control (No Intervention): Supervisors in the business-as-usual waitlist control condition will supervise teachers as-per-usual (i.e., using standard administrative supervision), and will be eligible for the typical array of professional development opportunities that may be offered to them. These supervisors will receive the Reflective Supervision enhancement the following academic year.

INTERVENTIONS:
Behavioral: Reflective Supervision Enhancement — The Reflective Supervision enhancement is a professional development series designed to train and support directors and education coordinators supervising state pre-kindergarten classrooms in using a reflective supervision approach with their staff.
  Arms: Reflective Supervision Enhancement

SUMMARY:
The goal of this clinical trial is to test an enhancement to early care and education, which is a professional development series that includes a foundational training and skill development workshops focused on training and supporting early learning supervisors in Reflective Practice and Supervision. Directors and education coordinators within state pre-kindergarten programs, and the teachers they supervise, will be the focus of this research. Hypothesized outcomes include promotion of reflective capacity and supervisory skill in supervisors, more effective supervisor-supervisee interactions, increases in reflective functioning and well-being in supervisees, increases in positive teaching practices and observed classroom quality, and increases in adaptive social-emotional development among children alongside prevention of emotion regulation difficulties. Researchers will compare whether these outcomes differ between participants who are currently receiving the Reflective Supervision enhancement and participants who are in the waitlist control condition.

ELIGIBILITY:
Inclusion Criteria:

* Supervisor in Rhode Island state pre-kindergarten program

Exclusion Criteria:

* Does not meet inclusion criteria above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-05-18 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Teaching Progress Assessment at 9 months | At baseline (beginning of academic year), and in 9 months
  Rhode Island Department of Education record review
Change from Baseline Teaching Progress Assessment at 12 months | At baseline (beginning of academic year), and in 12 months
  Rhode Island Department of Education record review
Change from 9-month Teaching Progress Assessment at 12 months | At 9 months (end of academic year), and in 12 months (beginning of next academic year)
  Rhode Island Department of Education record review
Change from Baseline Observed Classroom Quality at 9 months | At baseline (beginning of academic year), and in 9 months
  Pre-K Classroom Assessment Scoring System, scores range from 1 (minimally characteristic) to 7 (highly characteristic), with higher scores indicating higher classroom quality
Change from Baseline Observed Classroom Quality at 12 months | At baseline (beginning of academic year), and in 12 months
  Pre-K Classroom Assessment Scoring System, scores range from 1 (minimally characteristic) to 7 (highly characteristic), with higher scores indicating higher classroom quality
Change from 9-month Observed Classroom Quality at 12 months | At 9 months (end of academic year), and in 12 months (beginning of next academic year)
  Pre-K Classroom Assessment Scoring System, scores range from 1 (minimally characteristic) to 7 (highly characteristic), with higher scores indicating higher classroom quality
Change from Baseline Child Social-Emotional Functioning as assessed by Cognitive Toybox at 9 months | At baseline (beginning of academic year), and in 9 months
  Rhode Island Department of Education record review
Change from Baseline Child Emotion Regulation at 9 months | At baseline (beginning of academic year), and in 9 months
  Social Competence Scale - Teacher Version, Emotion Regulation subscale, scores range from 0 to 4 with higher scores indicating greater emotion regulation
Change from Baseline Child Prosocial/Communication Skills at 9 months | At baseline (beginning of academic year), and in 9 months
  Social Competence Scale - Teacher Version, Prosocial/Communication subscale, scores range from 0 to 4 with higher scores indicating greater prosocial/communication skills
Change from Baseline Child Social Competence at 9 months | At baseline (beginning of academic year), and in 9 months
  Social Competence Scale - Teacher Version, Total Social Competence Score, scores range from 0 to 4 with higher scores indicating greater social competence
Change from Baseline Child-Teacher Relationship Quality at 9 months | At baseline (beginning of academic year) and in 9 months
  Student-Teacher Relationship Scale - Short Form, scores range from 1 to 5 with higher scores indicating a more positive relationship

SECONDARY OUTCOMES:
Change from Baseline Supervisor Reflective Capacity at 9 months | At baseline (beginning of academic year) and in 9 months
  Reflective Supervision Rating Scale, Adapted Version, scores range from 1 to 4 with higher scores indicating greater reflective capacity
Change from Baseline Supervisory Competence at 9 months | At baseline (beginning of academic year) and in 9 months
  Supervisor Self-Assessment, scores range from 1 to 5 with higher scores indicating greater supervisory competence
Change from Baseline Supervisor Reflective Functioning at 9 months | At baseline (beginning of academic year) and in 9 months
  Reflective Functioning Questionnaire, scores range from 1 to 7 with higher scores indicating greater reflective functioning
Change from Baseline Supervisor Well-Being at 9 months | At baseline (beginning of academic year) and in 9 months
  Professional Quality of Life Scale, scores range from 1 to 5 with higher scores indicating greater well-being
Change from Baseline Quality of Reflective Supervision Relationship at 9 months | At baseline (beginning of academic year) and in 9 months
  Reflective Interaction Observation Scale, scores range from 1 to 5 with higher scores indicating a higher quality relationship
Program Climate assessed by Early Childhood Environment Rating Scale-Revised | At 9 months (end of academic year)
  Rhode Island Department of Education record review
Change from Baseline Supervisor Reflective Capacity at 9 months assessed by teacher-report | At baseline (beginning of academic year) and in 9 months
  Reflective Supervision Rating Scale, scores range from 1 to 4 with higher scores indicating greater reflective capacity
Change from Baseline Teacher Reflective Functioning at 9 months | At baseline (beginning of academic year) and in 9 months
  Reflective Functioning Questionnaire, scores range from 1 to 7 with higher scores indicating greater reflective functioning
Change from Baseline Teacher Well-Being at 9 months | At baseline (beginning of academic year) and in 9 months
  Professional Quality of Life Scale, scores range from 1 to 5 with higher scores indicating greater well-being
Change from Baseline Child Academic Functioning as assessed by Cognitive Toybox at 9 months | At baseline (beginning of academic year) and in 9 months
  Rhode Island Department of Education record review
Change from Baseline Child Academic Skills at 9 months | At baseline (beginning of academic year) and in 9 months
  Social Competence Scale - Teacher Version, Academic Skills subscale, scores range from 0 to 4 with higher scores indicating greater academic skills

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay P Huffhines, PhD, Principal Investigator — Bradley Hospital
Locations (1):
- Bradley Hospital, Riverside, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Final datasets generated from questionnaire, record review, and observational assessments will be available upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Requests for de-identified datasets will be honored within 30 months following completion of the project or at the time of the publication of manuscripts that present the main aims of the study
Access Criteria: A public use de-identified dataset that does not include sensitive or potentially identifiable information will be made available upon reasonable request. For datasets that include sensitive or potentially identifiable information, data-use agreements will be put in place with appropriate restrictions prior to the provision of data.